CLINICAL TRIAL: NCT04883216
Title: Investigation of the Characteristics of Chronic Pain Developing After COVID-19 in Patients With COVID-19
Brief Title: Investigation of the Characteristics of Chronic Pain Developing After COVID-19
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mert Zure, Medical Doctor, Istanbul University
Other Study IDs: 2021/389
Record Dates: First submitted 2021-05-09; First posted 2021-05-12 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Covid19; Coronavirus; Chronic Pain
Keywords: Chronic Pain; COVID19; Characteristics
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Data on pain after COVID-19 were generally collected from hospitalized patients and only include information on acute pain conditions. However, the characteristics of the chronic pain experienced after COVID-19 are unknown. For this reason, the treatment and recommendations for patients who present with chronic pain after COVID-19 are not clear. Our goal is to determine the characteristics and risk factors of chronic pain developing in COVID-19 patients and to create specific treatment recommendations for these patient groups with further studies.

DETAILED DESCRIPTION:
Data on pain developing after COVID-19 were generally collected from hospitalized patients and only include information on acute pain conditions seen after the ilness. It is noteworthy that headache and musculoskeletal pain were seen common in first few weeks. However, the characteristics (mechanical, inflammatory, central sensitization, anxiety-related, etc.) of the chronic pain experienced are unknown. For this reason, the treatment and recommendations for patients who present with chronic pain after COVID-19 are not clear. Our goal is to determine the characteristics and risk factors of chronic pain developing in COVID-19 patients and to create specific treatment recommendations for these patient groups with further studies.

ELIGIBILITY:
Inclusion Criteria:

1. Being over the age of 18
2. SARS-CoV-2 infection demonstrated with the PCR test (testing date irrelevant)
3. Pain developed or increased after having COVID-19

Exclusion Criteria:

1. Mental retardation or mental status not eligible to answer the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1120 patients who had previously suffered from COVID-19 disease will be included in the study upon application to physical medicine and rehabilitation outpatient clinics with pain complaints developed after COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 776 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Self-Leeds Assessment of Neuropathic Symptoms & Signs (S-LANSS) Pain Score | up to 1 year
  The S-LANSS aims to identify pain of predominantly neuropathic origin, as distinct from nociceptive pain, without the need for clinical examination.
The Hospital Anxiety and Depression Scale (HADS) Score | up to 1 year
  The Hospital Anxiety and Depression Scale (HADS) is a self-assessment questionnaire that has been found to be a reliable instrument for detecting states of anxiety and depression in the setting of hospital outpatient clinic. The HADS questionnaire has seven items each for depression and anxiety subscales.
Central Sensitization Inventory (CSI) | up to 1 year
  The Central Sensitisation Inventory (CSI) is a self-report outcome measure designed to identify patients who have symptoms that may be related to central sensitisation (CS) or central sensitivity syndromes (CSS) such as fibromyalgia, neck injury, temporomandibular joint disorder or migraine/tension headaches. CSI includes 25 questions related to common CSS symptoms.
Self-report Demographic Questionnaire | up to 1 year
  A questionnaire made by the researchers to understand the demographic characteristics of the patients included.
Visual Analog Scale (VAS) for Pain | up to 1 year
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül Ketenci, Professor, Study Director — Professor; Mert Zure, Expert, Principal Investigator — MD
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weng LM, Su X, Wang XQ. Pain Symptoms in Patients with Coronavirus Disease (COVID-19): A Literature Review. J Pain Res. 2021 Jan 26;14:147-159. doi: 10.2147/JPR.S269206. eCollection 2021. PMID 33531833
- [Background] Brooks SK, Webster RK, Smith LE, Woodland L, Wessely S, Greenberg N, Rubin GJ. The psychological impact of quarantine and how to reduce it: rapid review of the evidence. Lancet. 2020 Mar 14;395(10227):912-920. doi: 10.1016/S0140-6736(20)30460-8. Epub 2020 Feb 26. PMID 32112714
- [Background] Ding Y, He L, Zhang Q, Huang Z, Che X, Hou J, Wang H, Shen H, Qiu L, Li Z, Geng J, Cai J, Han H, Li X, Kang W, Weng D, Liang P, Jiang S. Organ distribution of severe acute respiratory syndrome (SARS) associated coronavirus (SARS-CoV) in SARS patients: implications for pathogenesis and virus transmission pathways. J Pathol. 2004 Jun;203(2):622-30. doi: 10.1002/path.1560. PMID 15141376
- [Background] Eccles R. Understanding the symptoms of the common cold and influenza. Lancet Infect Dis. 2005 Nov;5(11):718-25. doi: 10.1016/S1473-3099(05)70270-X. PMID 16253889